CLINICAL TRIAL: NCT06600412
Title: Effects of the ABCA1 Inducer R3R01 on Albuminuria Levels in Diabetic Kidney Disease
Brief Title: The Evaluation of the Drug R3R01 for the Excretion of Protein in the Urine in Patients With Diabetic Kidney Disease.
Acronym: Kidney ABC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: River 3 Renal Corp. (Industry)
Collaborators: Region Hovedstadens Apotek (Other Government); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3R01-DKD-201
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- R3R01 (Experimental): R3R01 oral tablet (200 mg twice daily) for 12 weeks
  Interventions: Drug: R3R01
- Placebo (Placebo Comparator): Placebo oral tablet twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R3R01 — R3R01 is an ATP-binding cassette transporter A1 (ABCA1) inducer, which increases the efflux of cholesterol from the intracellular space in the kidney. Please refer to arm/group description for further information.
  Arms: R3R01
Drug: Placebo — Please refer to arm/group description for further information.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to to investigate whether the drug R3R01 has a beneficial effect on the amount of protein excreted in the urine in adult patients (above 18 years of age) with type 2 diabetes and resulting kidney disease.

The main questions it aims to answer are:

1. Does 3 months of treatment with 200mg of the drug R3R01 morning and evening have a beneficial effect on the amount of protein excreted in the urine in patients with type 2 diabetes and kidney disease?
2. Does R3R01 have an effect on kidney function and daily blood pressure?

Researchers will compare the results of 40 people who take R3R01 to 20 people who receive an inactive substance (placebo).

Participants will receive R3R01 or the placebo as an oral tablet and undergo a selection of medical examinations - such as:

* blood samples
* urine tests
* kidney tests involving a radiolabelled marker which is injected into the bloodstream and monitored via blood samples
* 24 hour blood pressure monitoring via a wearable device
* urine pregnancy test (if applicable)

DETAILED DESCRIPTION:
An increasing amount of evidence suggests that lipid dysmetabolism and accumulation in the kidneys play a central role in the pathogenesis of kidney disease. This lipotoxicity, in turn, may contribute to the development of albuminuria and chronic kidney disease.

One may surmise that interventions that reduce or prevent the progression of kidney lipid accumulation protect against the progression of kidney disease, including diabetic kidney disease (DKD). Therefore, it is possible inhibiting cholesterol absorption, might effectively protect against lipid accumulation and related disease in the kidneys.

R3R01 is an ATP-binding cassette transporter A1 (ABCA1) inducer, which increases the efflux of cholesterol from the intracellular space in the kidney.

Persons with type 2 diabetes with moderate and severe albuminuria have a poor renal and cardiovascular prognosis. As albuminuria is viewed both as a risk marker but also as a target for intervention, any treatment with antiproteinuric effects could be beneficial. The role of ABCA1 inducer treatment on kidney parameters in diabetic kidney disease is not known. By investigating the impact of ABCA1 inducer treatment on albuminuria, it will be determined whether this intervention may represent a future treatment option.

This study is a single center, double-blind, placebo controlled, parallel group randomized (2:1) study, in 60 people with type 2 diabetes with moderate or severe albuminuria and estimated glomerular filtration rate (eGFR) above 30 ml/min/1.73m2. 40 people will take R3R01 whilst 20 people receive the placebo.

The study's primary objective is to evaluate the effect of 12 weeks treatment with R3R01 on albuminuria in the study population. In addition to a 12 week treatment period, there will be a follow-up period of approximately 24 weeks (168 days). The expected total duration of study participation is up to 36 weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (above 18 years of age) with controlled type 2 diabetes (hemoglobin A1c less than 10.5%).
2. Stable antihypertensive treatment 4 weeks before start of study drug and throughout study duration.
3. Titrated to the maximal dose or maximal tolerated dose of renin-angiotensin blocking treatment.
4. Stable treatment with lipid lowering agents for at least 4 weeks.
5. People on SGLT2-Inhibitors should be on a stable dose of the drug for at least 3 months.
6. UACR >30 mg/g and < 5000 mg/g on two consecutive measurements.
7. eGFR >30 ml/min/1.73 m2 (CKD-EPIcrea formula).
8. Abdominal obesity Women: > 88 cm, Men: > 102 cm or fasting triglyceride >2.0 mmol/l.
9. Systolic blood pressure ≥110 mmHg and ≤160 mmHg.
10. Both female patients, as well as female partners of male patients who are of child-bearing potential must be willing to not become pregnant for the complete duration of the study and 90 days after the last dose of study medication.
11. Males (including sterilized subjects) whose female partners have child-bearing potential, must agree to use male contraception (condoms) during the period from the time of signing the informed consent form through 90 days after the last dose of study drug. They must agree to immediately inform the investigator if their partner becomes pregnant during the study.

Exclusion Criteria:

1. Polycystic kidney disease, ANCA-associated vasculitis, or lupus nephritis.
2. Ongoing cancer treatment.
3. Immunosuppressive therapy or immunosuppression the prior 6 months.
4. Nephrotic syndrome.
5. Impaired liver function (clinically significant).
6. Pregnancy or lactation.
7. Failure to understand patient information or to collaborate with the investigator.
8. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study unless they agree to use highly effective contraception.
9. History of hypersensitivity to study drug and/or any of its excipients.
10. Hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
11. Active or planned treatment with a medication that interacts with R3R01.
12. Any other medical condition(s) that might put the patient at risk or influence study results in the investigators opinion, or that the investigator deems unsuitable for the study including drug or alcohol abuse or psychiatric, behavioral, or cognitive disorders sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin-to-creatinine ratio (UACR) | 12 weeks (84 days)
  Urinary albumin-to-creatinine ratio (UACR) (Change from baseline to end of treatment at 12 weeks (84 days).

SECONDARY OUTCOMES:
Measured or Estimated Glomerular Filtration Rate | 12 weeks (84 days)
  Measured glomerular filtration rate (GFR) with plasma clearance of 99Tc-DTPA or eGFR measured with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation based on creatinine and/or cystatin C (change from baseline to end of treatment at 12 weeks (84 days)).
24 hours ambulatory blood pressure | 12 weeks (84 days)
  24 hours ambulatory blood pressure (change from baseline to end of treatment at 12 weeks (84 days)).
Plasma Pharmacokinetics | 24 weeks (168 days)
  R3R01 plasma concentrations will be measured to determine Maximum plasma concentration (Cmax)
Plasma Pharmacokinetics | 24 weeks (168 days)
  R3R01 plasma concentrations will be measured to determine minimum blood plasma concentration (Cmin)
Plasma Pharmacokinetics | 24 weeks (168 days)
  R3R01 plasma concentrations will be measured to determine the half-life (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, dr.med., Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No